CLINICAL TRIAL: NCT00475072
Title: An Open Label Study to Evaluate the Safety and Effect on Sustained Virological Response of PEGASYS Plus Ribavirin in Patients With Hemophilia A and Chronic Hepatitis C
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) Plus Ribavirin in Hemophiliac Patients With Chronic Hepatitis C.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML16814
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 48 weeks
Drug: ribavirin — 1000/1200mg po daily for 48 weeks

SUMMARY:
This study will evaluate the efficacy and safety of PEGASYS plus ribavirin in male patients with hemophilia A and chronic hepatitis C. All patients will receive PEGASYS 180 micrograms s.c. weekly plus ribavirin 1000-1200mg p.o. daily (depending on body weight) for 48 weeks. Following treatment there will be a 24 week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male patients, >=18 years of age;
* hemophilia A;
* chronic hepatitis C;
* compensated liver disease.

Exclusion Criteria:

* therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment <=6 months before start of study drug;
* hepatitis A, hepatitis B or HIV infection;
* chronic liver disease other than chronic hepatitis C.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
SVR | Week 72

SECONDARY OUTCOMES:
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Mexico City, Mexico